CLINICAL TRIAL: NCT00411905
Title: Phase I/II Study of Bortezomib and Low Dose Cytarabine in the Treatment of High-risk Myelodysplastic Syndromes
Brief Title: Bortezomib and Low Dose Cytarabine in the Treatment of High-risk Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Groupe Francophone des Myelodysplasies (Other)
Collaborators: Johnson & Johnson (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GFM BAR-C-2005
Record Dates: First submitted 2006-12-14; First posted 2006-12-15 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2010-07

CONDITIONS: Myelodysplastic Syndromes
Keywords: Myelodysplastic syndromes; IPSS Int-2 and High risk; Bortezomib; Low dose Cytarabine; Bone Marrow diseases
MeSH Terms: conditions — Myelodysplastic Syndromes; Bone Marrow Diseases | interventions — Bortezomib

STUDY DESIGN:
Intervention Model Description: Essai ouvert multicentrique de phase I-II
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Bortezomib

SUMMARY:
We are evaluating the efficacy of the association of Low dose Cytarabine in association with Bortezomib in the treatment of patients diagnosed with high risk Myelodysplastic syndromes. Our aim is to decrease transfusion requirements and if possible induce a complete or at least a partial remission.

DETAILED DESCRIPTION:
Four cycles of treatment are proposed at 28 day intervals in an ambulatory setting

Cycle 1 :

* Cytarabine 10 mg /m2/day subcutaneous injection for 14 days
* Bortézomib 1,5mg/m2 days 1,4,8,11

Cycles 2, 3, 4 :

* Cytarabine 20 mg /m2/j subcutaneous injections for 14 days
* Bortézomib 1,5mg/m2 days 1,4,8,11

Bone marrow aspirates are evaluated just before the first cycle, after the second and after the fourth cycles

Responding patients may continue the treatment for 2 further cycles

ELIGIBILITY:
Inclusion Criteria:

* MDS with IPSS scores Int-2 or High
* Life expectancy greater than 6 months
* No other available treatment options

Exclusion Criteria:

* MDS with IPSS scores Low or Int-1
* > 30% bone marrow blasts
* clinical neuropathy of greater than grade 2
* ECOG Score 3 or 4
* Creatinine clearance of < 30 ml/min
* LMMC
* Pregnant patients or lactating mothers
* Patients having received intensive chemotherapy in the 3 months prior to inclusion
* Patients with uncontrolled pulmonary, cardiac, neurological, gastro-intestinal or genito-urinary disorders

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2010-07-08 (Actual); Study Completion 2011-08-01 (Actual)

PRIMARY OUTCOMES:
Complete Response
Partial Response
Efficacy and safety evaluation | 18 mois
  A total of 138 cycles were administered. The median number of cycles administered was 3·2 (range 0·5-8). Thirty-six patients (84%) received at least two cycles and 17 (40%) received the planned four cycles, six responding patients received 1-4 additional cycles. Treatment was dis- continued in the responding patients at progression to AML or for toxicity.
  The most common treatment-related adverse events were related to myelosuppression . Neutropenia (Grade 4) and thrombocytopenia (Grade 4) were seen during treatment in 51% and 46% of the patients, respectively. Three of the patients with pre-treatment Grade 0-2 neutropenia and thrombocytopenia developed Grade 3-4 toxicity complicated by infection and bleeding. Grade 3-4 neutropenia was responsible for infection in six patients. Grade 3-4

SECONDARY OUTCOMES:
Hematological Improvement

CONTACTS AND LOCATIONS:
Overall Officials: Francois DREYFUS, MD PhD, Principal Investigator — Groupe francaise des Myelodysplasies
Locations (15):
- France (15):
  - CHU Angers, Angers
  - Hopital Avicenne, Bobigny
  - Institut Bergonie, Bordeaux
  - CHU de Caen, Caen
  - CHU Dijon, Dijon
  - CHU Albert Michallon, Grenoble
  - CHU de Limoges, Limoges
  - Hopital Paoli Calmette, Marseille
  - CHU Archet, Nice
  - Hopital Cochin, Paris
  - Centre Hospitalier Joffre, Perpignan
  - Centre Henry Becquerel, Rouen
  - Centre Hospitalier Universitaire de STRASBOURG, Strasbourg
  - CHU Purpan, Toulouse
  - CHU Brabois, Vandœuvre-lès-Nancy